CLINICAL TRIAL: NCT04889339
Title: Validation of a New Generation of Orthopedic Brace for Treating Adolescent Idiopathic Scoliosis by Using Growth Modulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Hubert Labelle, MD, Orthopedist, researcher, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-3437
Record Dates: First submitted 2021-05-03; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Scoliosis; Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Spine deformity; Brace; Growth modulation
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: The study will be separated into two stages. Each patient will initially try a control brace and a test brace in a crossover study model to evaluate the immediate correction. Each patient will then use one brace from either the control arm or test arm to evaluate the long-term correction of the brace.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group: Braces designed with growth modulation simulation (Experimental): The braces will be designed using a growth modulation method.
  Interventions: Device: Test brace versus control brace: Immediate correction; Device: Test brace versus control brace: Long-term correction
- Control group: Conventional method (Active Comparator): The braces will be designed by an orthotist without growth modulation simulation.
  Interventions: Device: Test brace versus control brace: Immediate correction; Device: Test brace versus control brace: Long-term correction

INTERVENTIONS:
Device: Test brace versus control brace: Immediate correction — The trunk surface will be scanned to reconstruct a numerical model of the patient's trunk, this reconstruction will help to produce the optimized brace. The patient skeletal will also be reconstructed from a bilateral radiograph using an EOS imaging system. Each patient will try both the control and the test brace. Radiographic and patient-reported data will be gathered and analyzed to observe changes between the immediate correction of the braces. The SRS-22r will be collected. The study protocol requires no additional visits beyond the standard of care. There will be one additional radiograph compared to the standard of care.
Device: Test brace versus control brace: Long-term correction — After comparing the immediate correction of the braces, each patient will be using either the test or the control brace for a period of two years. There will be follow-up visits, between 6 months and 1 year depending on the patient growth. The brace will be renewed using the same procedure to adapt to the patient's growth. The study protocol requires no additional visits beyond the standard of care. There will be no additional radiograph compared to the standard of care. Compliance monitors are installed in each brace.

SUMMARY:
Adolescent Idiopathic Scoliosis affects 3-4% of the Canadian population, of which about 10% will need a brace treatment during pubertal growth spurt. Our team has developed an innovative conception method for brace design by simulating the growth modulation using numerical models. Those models are customized to each patient. In this project, the investigators will evaluate the effectiveness of this platform customized treatment and validate its clinical application.

ELIGIBILITY:
Inclusion Criteria:

* AIS diagnosis
* Risser 0-2
* Primary curve angles 20 degrees - 40 degrees
* If female, either premenarchal or less than 18 months postmenarchal.

Exclusion Criteria:

* Patients with a pre-existing cardiovascular condition
* Patients with a symptom of a neurological disorder
* Patients with any other disorder of the musculoskeletal system affecting the lower limbs

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cobb angle | Baseline - 2 years
  Radiographics will be gathered and analyzed to observe changes between time points. All radiographs will be taken with an low-dose biplane radiographic system (EOS) to allow 3D reconstructions.

SECONDARY OUTCOMES:
Treatment failure rate | Baseline, 2 years
  Treatment failure is defined as having a Cobb angle progress by more than 5 degrees compared to the baseline measurement or exceeding a value of 45 degrees
Quality of Life (QoL) | Baseline, 2 years
  The QoL will be measured using the SRS-22r and MOBI questionnaire.
Immediate in-brace Cobb angle | 5 minutes after brace fitting
  Radiographics will be gathered and analyzed to observe changes between the control and test braces. All radiographs will be taken with an low-dose biplane radiographic system (EOS).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada